CLINICAL TRIAL: NCT00837824
Title: A Phase 2, Randomized, Open Label, Dose-Ranging, Multiple Dose Study of Fabrazyme® In Patients With Fabry Disease and With Severe Renal Disease
Brief Title: Severe Renal Disease Study in Fabry Patients Treated With Fabrazyme
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated early due to inadequate study design.
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: CRL/Medinet (Unknown)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGAL-022-02
Record Dates: First submitted 2008-10-23; First posted 2009-02-05 (Estimated); Results first posted 2009-02-05 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Fabry Disease; Chronic Kidney Disease, Stage IV (Severe)
Keywords: Fabry Disease patients with Severe Renal Disease
MeSH Terms: conditions — Fabry Disease; Renal Insufficiency, Chronic | interventions — agalsidase beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fabrazyme 1mg/kg every 2 weeks (Experimental): Fabrazyme 1.0 mg/kg every 2 weeks
  Interventions: Biological: Fabrazyme (agalsidase beta)
- Fabrazyme 3mg/kg every 2 weeks (Experimental): Fabrazyme 3.0 mg/kg every 2 weeks
  Interventions: Biological: Fabrazyme (agalsidase beta)

INTERVENTIONS:
Biological: Fabrazyme (agalsidase beta) — 1.0 mg/kg every 2 weeks
  Other Names: r-hαGAL
  Arms: Fabrazyme 1mg/kg every 2 weeks
Biological: Fabrazyme (agalsidase beta) — 3.0 mg/kg every 2 weeks
  Other Names: r-hαGAL
  Arms: Fabrazyme 3mg/kg every 2 weeks

SUMMARY:
This study was designed to determine appropriate treatment with Fabrazyme at a biweekly dose of either 1 mg/kg or 3 mg/kg in a population of patients with severe renal disease burden.

ELIGIBILITY:
Inclusion Criteria:

* provided written informed consent prior to any study-related procedures being performed.
* be ≥16 years old.
* have a current diagnosis of Fabry disease (defined as abnormal α-galactosidase (α GAL) enzyme levels or Fabry genotype).
* have one of the following clinical conditions present at enrollment: serum creatinine level greater than 3.0 mg/dL (an average of two values at least one week apart), or be currently on dialysis, or be status post kidney transplant by greater than 3 months.
* have the ability to comply with the requirements of the protocol
* have a negative pregnancy test, if a female patient of childbearing potential. In addition, all female patients of childbearing potential must use a medically accepted method of contraception throughout the study.

Exclusion Criteria:

* if they did not meet the specific inclusion criteria.
* if they had participated in a study employing an investigational drug within 30 days of the start of their participation in this trial.
* had previously received enzyme replacement therapy (ERT) for their Fabry disease.
* had diabetic nephropathy.
* were pregnant or lactating.
* were unwilling to comply with the requirements of the protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-12; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (9):
- United States (9):
  - Farmington, Connecticut
  - Coral Springs, Florida
  - Kansas City, Kansas
  - Boston, Massachusetts
  - New York, New York
  - Rochester, New York
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Because the study was ended early only 20 patients from 9 sites were randomized into this study using a 1:1 randomization scheme to receive biweekly infusions of either 1 mg/kg (11 patients) or 3 mg/kg (9 patients) of Fabrazyme.
Period: Overall Study
Arm/Group | Fabrazyme 1mg/kg Every 2 Weeks | Fabrazyme 3mg/kg Every 2 Weeks
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fabrazyme 1mg/kg Every 2 Weeks | Fabrazyme 3mg/kg Every 2 Weeks | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Customized [Number; unit: Years]
  < 40 Years | 1 | 1 | 2
  ≥ 40 Years | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (6.96) | 48.9 (7.55) | 49.2 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 10 | 7 | 17
Race/Ethnicity, Customized [Number; unit: Number of Participants]
  Caucasian | 7 | 7 | 14
  Black | 3 | 2 | 5
  Hispanic | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinically Significant Progression of Cardiac Disease, Cerebrovascular Disease, and/or Death Among Fabry Patients With Severe Kidney Disease
Description: The trial was terminated early due to inadequate study design. During the study period of 7 months, only 1 patient had a clinical event, a stroke, in the Fabrazyme 1 mg/kg treatment arm. The time to event was determined from first dose of Fabrazyme to the date of event.
Time Frame: 7 months
Population: Intent-to-Treat (ITT) Population-consisted of all 20 patients enrolled in the trial. The original sample size was 120 patients. Due to early termination, only 20 patients were enrolled in this trial. No imputation of data was performed. During the 7 months study period, only 1 patient had a clinical event in the Fabrazyme 1 mg/kg treatment arm.
Measure: Number; unit: Days
Arm/Group | Fabrazyme 1mg/kg Every 2 Weeks | Fabrazyme 3mg/kg Every 2 Weeks
Number analyzed (Participants) | 1 | 0
Days | 35 |

2. Secondary Outcome: Plasma Globotriaosylceramide (GL-3)
Description: This outcome measure evaluated the mean plasma GL-3 values for all patients to see if it decreased while on Fabrazyme. Normal plasma GL-3 level is defined as ≤ 7.03 µg/mL.
Time Frame: Evaluated at Baseline, Month 3, and Final Visit
Population: Fabrazyme 1mg/kg every 2 weeks: ITT population - 11 patients at baseline, 7 patients at Month 3, and 9 patients at Final Visit had Plasma GL-3 values.
  Fabrazyme 3mg/kg every 2 weeks: ITT population - 9 patients at baseline, 2 patients at Month 3, and 7 patients at Final Visit had Plasma GL-3 values
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Fabrazyme 1mg/kg Every 2 Weeks | Fabrazyme 3mg/kg Every 2 Weeks
Number analyzed (Participants) | 11 | 9
µg/mL
  Plasma GL-3 at Baseline | 8.7 (3.33) | 8.3 (3.92)
  Plasma GL-3 at Month 3 | 5.1 (2.05) | 5.6 (0.28)
  Plasma GL-3 at Final Visit | 5.1 (1.53) | 4.9 (1.74)

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Fabrazyme 1mg/kg Every 2 Weeks | Fabrazyme 3mg/kg Every 2 Weeks | Total
Serious Adverse Events (participants affected / at risk) | 4/11 | 1/9 | 5/20
Other Adverse Events (participants affected / at risk) | 10/11 | 9/9 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fabrazyme 1mg/kg Every 2 Weeks (N=11) | Fabrazyme 3mg/kg Every 2 Weeks (N=9) | Total (N=20)
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fabrazyme 1mg/kg Every 2 Weeks (N=11) | Fabrazyme 3mg/kg Every 2 Weeks (N=9) | Total (N=20)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Adverse event (General disorders) | 1 | 0 | 1
Chills (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 1 | 2
Feeling hot (General disorders) | 1 | 0 | 1
Influenza like illness (General disorders) | 1 | 1 | 2
Malaise (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 3 | 3
Pain (General disorders) | 1 | 1 | 2
Pyrexia (General disorders) | 2 | 0 | 2
Sluggishness (General disorders) | 1 | 0 | 1
Arteriovenous fistula site infection (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 1 | 1
Blood calcium decreased (Investigations) | 0 | 1 | 1
Blood phosphorus increased (Investigations) | 0 | 1 | 1
Breath sounds abnormal (Investigations) | 0 | 1 | 1
Haematocrit decreased (Investigations) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 1
Red blood cell count decreased (Investigations) | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 3
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
The trial was terminated early due to inadequate study design, leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.